CLINICAL TRIAL: NCT06595641
Title: Effect of Transfer Energy Capacitive Resistive Therapy on Shoulder Pain and Function in Shoulder Impingement Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mahmoud Abdelaziz Khalil, Director, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005345
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Impingement Syndrome, Shoulder
Keywords: Strengthening Exercises; Shoulder Impingement Syndrome; Transfer energy capacitive and resistive
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- strength training program group (Active Comparator): In Group I, fifteen patients will undergo a 3-week exercise program, with sessions lasting 35-45 minutes, three times a week. Each session includes five exercises, each performed for three sets of 10 repetitions:
  Shoulder Retraction - Strengthens muscles between shoulder blades. Shoulder Scaption - Improves stability and range of motion. Shoulder External Rotation from Side Lying - Targets rotator cuff muscles. Shoulder Protraction - Enhances shoulder blade function. Shoulder Extension - Strengthens posterior shoulder muscles.
  Interventions: Other: strength training program
- Experimental TECAR Group (Experimental): In the experimental group, fifteen patients will follow a three-week program that combines targeted exercises with Transfer Energy Capacitive and Resistive (TECAR) therapy. Each session of the exercise program, conducted three times a week, will include a series of five shoulder exercises: retraction, scaption, external rotation from a side-lying position, protraction, and extension.
  Alongside these exercises, patients will receive TECAR therapy, which involves applying high-frequency electromagnetic energy to the affected shoulder. During the therapy, a capacitive electrode will first be used for ten minutes to target the soft tissues near the biceps. Following this, the therapy will switch to the resistive mode for another ten minutes, focusing on the deeper tissues around the T1-T9 vertebrae. Each TECAR session will last for a total of twenty minutes, and patients will undergo this treatment nine times over the course of the study, with three sessions each week.
  Interventions: Device: Transfer Energy Capacitive Resistive Therapy; Other: strength training program

INTERVENTIONS:
Device: Transfer Energy Capacitive Resistive Therapy — It's a physical treatment modality commonly used to treat musculoskeletal pain. It normally uses a longwave radiofrequency of ~0.5 MHz. The system consists of a neutral plate and two different electrodes that can transfer energy in two modalities: capacitive and resistive
  Other Names: TECAR
  Arms: Experimental TECAR Group
Other: strength training program — Each session includes five exercises, each performed for three sets of 10 repetitions:
  Shoulder Retraction - Strengthens muscles between shoulder blades. Shoulder Scaption - Improves stability and range of motion. Shoulder External Rotation from Side Lying - Targets rotator cuff muscles. Shoulder Protraction - Enhances shoulder blade function. Shoulder Extension - Strengthens posterior shoulder muscles

SUMMARY:
This study investigates the efficacy of combining Transfer Energy Capacitive and Resistive (TECAR) therapy with standard strengthening exercises in treating Shoulder Impingement Syndrome (SIS). A double-blinded randomized controlled trial will compare outcomes between patients receiving only strengthening exercises and those receiving both TECAR therapy and exercises. Key outcomes include improvements in pain, muscle strength, joint position sense, and shoulder function. The study aims to determine if TECAR therapy enhances treatment benefits beyond those achieved with exercises alone.

DETAILED DESCRIPTION:
Background: Shoulder Impingement Syndrome (SIS) is a prevalent musculoskeletal condition characterized by pain and functional impairment due to the compression of rotator cuff tendons beneath the coracoacromial arch. Despite the effectiveness of conservative treatments such as strengthening exercises, there is emerging interest in additional modalities, including Transfer Energy Capacitive and Resistive (TECAR) therapy. TECAR therapy utilizes high-frequency electromagnetic waves to provide deep thermal energy, potentially enhancing tissue repair and pain relief.

Objective: This study aims to evaluate the effectiveness of combining TECAR therapy with a standard strengthening exercise regimen compared to strengthening exercises alone in patients with SIS.

Methods: A double-blinded randomized controlled trial will be conducted with 30 participants diagnosed with Neer's Stage I SIS. Participants will be randomly assigned to either a control group receiving only strengthening exercises or an experimental group receiving both TECAR therapy and strengthening exercises. The study will assess pain, shoulder muscle strength, joint position sense, and shoulder function using a range of validated instruments including the Visual Analogue Scale (VAS), Hand-Held Dynamometer (HHD), Digital Inclinometer, and the Shoulder Pain and Disability Index (SPADI).

ELIGIBILITY:
Inclusion Criteria:

* Both gender age from 25-40 with a clinical diagnosis of Neer's stage II SIS and body mass index (18.5-29.9)

  * Shoulder pain for at least three months
  * Painful arc of movement during flexion or abduction
  * Positive Neer's or kennedy- hawkins test or empty can test
  * Pain on resisted external rotation, abduction

Exclusion Criteria:

* Symptoms of cervical radiculopathy.

  * Diagnosed inflammatory disorder.
  * Neurological disorder.
  * Widespread pain condition.
  * Evidence of complete rotator cuff tear (positive drop arm test).
  * Previous surgery to the affected shoulder.
  * Noncompliance patient.
  * Pacemaker.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 3 weeks
  which rates pain intensity from 0 (no pain) to 10 (worst possible pain)

SECONDARY OUTCOMES:
Manual Muscle Test System (MMT) | 3 weeks
  will be used to obtain normative strength values for both external and internal shoulder rotators .
Joint Position Sense of the Shoulder joint | 3 weeks
  All participants will be submitted to the evaluation of the JPS at 30° and 120° of shoulder forward flexion, using a digital inclinometer
shoulder Function Using the Arabic SPADI Questionnaire | 3 weeks
  The Arabic SPADI is recommended for the evaluation of Arabic-speaking patients with shoulder dysfunction . To answer the questions, patients will be asked to place a mark on a 10 cm visual analogue scale for each question. Verbal anchors for the pain dimension are 'no pain at all' and 'worst pain imaginable', and those for the functional activities are 'no difficulty' and 'so difficult, it required help'. The scores from both dimensions are averaged to derive a total score

CONTACTS AND LOCATIONS:
Overall Officials: Enas Fawzy Youssif, Professor, Study Chair — Cairo University; ahmed mohamed khalil, PhD, Study Director — Pharos University in Alexandria; Sherif Hamdy Zawam, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Davies H, Wells F, Czarkowski M. Standards for research ethics committees: purpose, problems and the possibilities of other approaches. J Med Ethics. 2009 Jun;35(6):382-3. doi: 10.1136/jme.2008.027722. PMID 19482984
- [Result] Yi SD, Baek SK. Interrupted coarsening in the zero-temperature kinetic Ising chain driven by a periodic external field. Phys Rev E Stat Nonlin Soft Matter Phys. 2015 Jun;91(6):062107. doi: 10.1103/PhysRevE.91.062107. Epub 2015 Jun 5. PMID 26172661
- [Result] Braun BJ, Osche D, Rollmann M, Orth M, Morsdorf P, Histing T, Pohlemann T, Herath SC. Increased therapy demand and impending loss of previous residence status after proximal femur fractures can be determined by continuous gait analysis - A clinical feasibility study. Injury. 2019 Jul;50(7):1329-1332. doi: 10.1016/j.injury.2019.05.007. Epub 2019 May 18. PMID 31178148
- See also: The Effectiveness of an Upper Extremity Neuromuscular Training Program on the Shoulder Function of Military Members With a Rotator Cuff Tendinopathy: A Pilot Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/31178148
- See also: Effectiveness of microwave diathermy on pain, functional capacity, muscle strength, quality of life, and depression in patients with subacromial impingement syndrome: a randomized placebo-controlled clinical study — https://pubmed.ncbi.nlm.nih.gov/26172661
- See also: Restricted scapular mobility during arm abduction: implications for impingement syndrome — https://pubmed.ncbi.nlm.nih.gov/19482984